CLINICAL TRIAL: NCT05920746
Title: Type of Magnetic Field and the Effects of Rheumatoid Arthritis Treatment
Brief Title: Treatment of Rheumatoid Hand With Magnetotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jolanta Zwolińska (Other)
Responsible Party: Sponsor-Investigator, Jolanta Zwolińska, Doctor of Philosophy, University of Rzeszow
Organization: University of Rzeszow (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Universyty of Rzeszow
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Rheumatoid Arthritis; Hand Rheumatism
Keywords: Magnetotherapy; Rheumatoid arthritis; Hand function
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Magnetic Field Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Assessor evaluating the patients' condition had no knowledge of the outcome of randomization of patients to the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotherapy with Static Magnetic Field (Experimental): Patients have kinesiotherapy of hand and static magnetic field. All patients without steroid anti-inflammatory drugs.
  Interventions: Other: Kinesiotherapy with magnetotherapy
- Kinesiotherapy with low-frequency pulsed magnetic field (Experimental): Patients have kinesiotherapy of hand and low-frequency pulsed magnetic field. All patients without steroid anti-inflammatory drugs.
  Interventions: Other: Kinesiotherapy with magnetotherapy

INTERVENTIONS:
Other: Kinesiotherapy with magnetotherapy — Individual kinesiotherapy. Parameters of magnetic field: 7 mT, f= 10-20 Hz, type of impulse: bipolar, rectangular pulse
  Other Names: Kinesiotherapy with static magnetic field; Kinesiotherapy with low-frequency pulsed magnetic field

SUMMARY:
Brief Summary:

Participants with rheumatoid arthritis with recommendation to physiotherapy.

Created 2 study groups:

1. Kinesiotherapy with static magnetic field
2. Kinesiotherapy with low-frequency pulsed magnetic field

Pulsed magnetic field give better effects then static magnetic field.

DETAILED DESCRIPTION:
Participants with rheumatoid arthritis with recommendation to physiotherapy. All participants have dysfunction and pain of hand. Before entering the study, all patients were examined by a rheumatologist, who determined the degree of radiological and functional changes and measured blood pressure. Patients with II° and III° of radiological and functional changes were qualified for the study. All the patients gave their informed consent to participate in the study. The examination included an overall assessment of functional status. Patients were examined immediately before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Informed voluntary consent to participate in the study
2. II ° and III ° of advancement of radiological changes
3. II ° and III ° of advancement of functional changes
4. Remission, low or moderate RA activity: DAS28
5. Medical referral for physiotherapy treatment

Exclusion Criteria:

1. Additional physiotherapy treatments for the hands
2. Contraindications for magnetotherapy treatments
3. Lack of informed, voluntary consent to participate in the study

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Change from baseline VAS value immediately after therapy.
  Pain severity rating scale. only one value. Minimum value is 0, maximum value is 10. The best is 0, the worst is 10.
Health Assesment Questionaire | Change from baseline HAQ-20 value immediately after therapy.
  Subjective assesment of level of disability. Value of each of 8 subsections: minimum value 0, maximum value 3. total score is averaged. The best total score is 0, the worst is 3.
Range of motion | Change from baseline range of motion value immediately after therapy.
  Computerized measurement of the range of motion of the joints of the hand [mm]. A higher score value meant a greater range of motions.
Displacement hand volume measurement | Change from baseline volume value immediately after therapy.
  Measurement of hand volume using the displacement method [mm3]. The higher score means less swelling.
Persistence time of morning stiffness | Change from baseline time of morning stiffness value immediately after therapy.
  Patient's subjective assessment of the duration of morning stiffness [min]. The longer durations means more hand dysfunction.
Severity of morning stiffness | Change from baseline time of severity of morning stiffness value immediately after therapy.
  Assessing the severity of morning stiffness using a 100-point scale. The higher score means a greater severity of morning stiffness.

CONTACTS AND LOCATIONS:
Overall Officials: Jolanta Zwolinska, PhD, Principal Investigator — University of Rzeszow
Locations (1):
- Laboratorium Czynników Fizykalnych w Rehabilitacji w Przyrodniczo-Medycznym Centrum Badań Innowacyjnych Uniwersytetu Rzeszowskiego, Rzeszów, Podkarpackie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parate D, Franco-Obregon A, Frohlich J, Beyer C, Abbas AA, Kamarul T, Hui JHP, Yang Z. Enhancement of mesenchymal stem cell chondrogenesis with short-term low intensity pulsed electromagnetic fields. Sci Rep. 2017 Aug 25;7(1):9421. doi: 10.1038/s41598-017-09892-w. PMID 28842627
- [Result] Tong J, Chen Z, Sun G, Zhou J, Zeng Y, Zhong P, Deng C, Chen X, Liu L, Wang S, Chen J, Liao Y. The Efficacy of Pulsed Electromagnetic Fields on Pain, Stiffness, and Physical Function in Osteoarthritis: A Systematic Review and Meta-Analysis. Pain Res Manag. 2022 May 9;2022:9939891. doi: 10.1155/2022/9939891. eCollection 2022. PMID 35586276
- [Result] Chen Y, Aspera-Werz RH, Menger MM, Falldorf K, Ronniger M, Stacke C, Histing T, Nussler AK, Ehnert S. Exposure to 16 Hz Pulsed Electromagnetic Fields Protect the Structural Integrity of Primary Cilia and Associated TGF-beta Signaling in Osteoprogenitor Cells Harmed by Cigarette Smoke. Int J Mol Sci. 2021 Jun 29;22(13):7036. doi: 10.3390/ijms22137036. PMID 34210094
- [Result] Dundar U, Asik G, Ulasli AM, Sinici S, Yaman F, Solak O, Toktas H, Eroglu S. Assessment of pulsed electromagnetic field therapy with Serum YKL-40 and ultrasonography in patients with knee osteoarthritis. Int J Rheum Dis. 2016 Mar;19(3):287-93. doi: 10.1111/1756-185X.12565. Epub 2015 May 8. PMID 25955771
- [Result] Wu Z, Ding X, Lei G, Zeng C, Wei J, Li J, Li H, Yang T, Cui Y, Xiong Y, Wang Y, Xie D. Efficacy and safety of the pulsed electromagnetic field in osteoarthritis: a meta-analysis. BMJ Open. 2018 Dec 14;8(12):e022879. doi: 10.1136/bmjopen-2018-022879. PMID 30552258